CLINICAL TRIAL: NCT05665244
Title: To Determine the Efficacy of Topical Cryotherapy on Supraglottic Laryngeal Mucosa in the Treatment of Chronic Neurogenic Cough in Adult Patients
Brief Title: Laryngeal Cryotherapy for Refractory Neurogenic Cough
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Shumon Dhar, MD, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0644
Record Dates: First submitted 2022-12-01; First posted 2022-12-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Upper-Airway Cough Syndrome
MeSH Terms: conditions — upper airway cough syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Upper airway cough syndrome
  Interventions: Procedure: Laryngeal cryotherapy; Device: Cryoprobe

INTERVENTIONS:
Procedure: Laryngeal cryotherapy — Laryngeal cryotherapy is the therapeutic freezing of tissue in the throat to numb the overactive sensory nerves in the throat. This technique is believed to reduce cough symptoms in this study.
Device: Cryoprobe — Cryoprobe is FDA approved for use for the destruction of unwanted tissue along the respiratory tract

SUMMARY:
This study aims to evaluate the safety and efficacy of upper aerodigestive tract cryotherapy treatment in patients with refractory neurogenic cough in a prospective pilot study with a validated patient reported outcome measure

DETAILED DESCRIPTION:
This study aims to test a new type of treatment for patients suffering from chronic cough, also known as upper airway cough syndrome. The new treatment involves the use of laryngeal cryotherapy which is the therapeutic freezing of tissue in the throat to numb the overactive sensory nerves in the throat which is believed to reduce cough symptoms. Patients will first undergo a flexible scope of the throat (laryngoscopy) to test for hypersensitive areas in the throat, then undergo the cryotherapy procedure in the office. After that, patients will be followed up in the clinic with the usual standard of care visits and undergo validated cough surveys to track their cough symptoms after the procedure. Possible side effects to this procedure are listed in detail below, and include temporary throat pain and coughing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years or older with diagnosis of neurogenic cough
* Neurogenic cough is a diagnosis of exclusion applied to persistent cough (8 weeks or longer)
* Negative workup for other causes, including sinonasal allergies/chronic sinusitis, cough-variant asthma, and GERD
* Patient willing to participate in a clinical trial

Exclusion Criteria:

* Uncontrolled reflux (scoring on Reflux Symptom index of 13 or higher)
* Vocal fold abnormalities or impairment
* History of asthma or other underlying lung condition not adequately treated or controlled
* Uncontrolled Allergic Rhinitis (Total Nasal Symptom Score >6, which would indicate moderate disease32)
* Reported symptom of postnasal drip
* Current smoker
* Current neuromodulator medication use
* Patient unwilling to participate in clinical trial or sign an informed consent
* End stage medical disease with poor life expectancy
* Medical instability deemed by the investigators as a contraindication for enrollment
* Abnormal Chest X-ray
* Abnormal pulmonary function testing (PFTs)
* Positive local allergy panel (combined RAST testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patient with eurogenic cough is a diagnosis of exclusion applied to persistent cough (8 weeks or longer) and of the age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Improved quality of life of patients suffering from chronic cough | 2 years
  This is a validated patient reported outcome measure for chronic cough. This is a questionnaire of 10 questions about cough symptoms, each question is rated on a scale of 0-4 by the patient. The higher the CSI total score the worsen the cough symptoms are for the patient. The CSI will be compared across 5 time points (Pre-Laryngeal Cryotherapy, 1 week post cryotherapy, 1 month post cryotherapy, 3 months post cryotherapy and 6 months post cryotherapy) using repeated measures one-way ANOVA. Post-hoc pair-wise comparisons with Bonferroni correction will be used, as appropriate.
Pre and Post-time point differences. | 2 years
  Sample size of 25 was determined based on expectations of a detectable significant within-group using a repeated measures ANOVA across 5 time points (add in the time points) with an alpha level of 0.0125, 85% power, and 1.246 effect size (based on previous work by Simpson et al PMID: 29668037.) needed to observe pre-post time point differences.

SECONDARY OUTCOMES:
Pre- and post-treatment measures for the cryotherapy treatment group | 2 years
  This measure is the pre cryotherapy and 1 week post cryotherapy laryngeal aesthesiometer testing. This is a type of validated sensory testing of the larynx performed during an office flexible laryngoscopy where calibrated monofilaments are used to assess how sensitive certain parts of the larynx are. The data collected will be if a specific monofilament (size 6-0, 5-0, and 4-0) can trigger or not trigger a cough reflex when applied to specific subsites of the larynx (aryepiglottic fold, laryngeal aspect of epiglottis, false vocal fold, arytenoid prominence, and lateral and medial piriform sinus

CONTACTS AND LOCATIONS:
Overall Officials: Shumon Dhar, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson CB, Amin MR. Chronic cough: state-of-the-art review. Otolaryngol Head Neck Surg. 2006 Apr;134(4):693-700. doi: 10.1016/j.otohns.2005.11.014. PMID 16564398
- [Background] Gibson P, Wang G, McGarvey L, Vertigan AE, Altman KW, Birring SS; CHEST Expert Cough Panel. Treatment of Unexplained Chronic Cough: CHEST Guideline and Expert Panel Report. Chest. 2016 Jan;149(1):27-44. doi: 10.1378/chest.15-1496. Epub 2016 Jan 6. PMID 26426314
- [Background] Farooqi MAM, Cheng V, Wahab M, Shahid I, O'Byrne PM, Satia I. Investigations and management of chronic cough: a 2020 update from the European Respiratory Society Chronic Cough Task Force. Pol Arch Intern Med. 2020 Sep 30;130(9):789-795. doi: 10.20452/pamw.15484. Epub 2020 Jul 6. PMID 32627514
- [Background] Simpson CB, Tibbetts KM, Loochtan MJ, Dominguez LM. Treatment of chronic neurogenic cough with in-office superior laryngeal nerve block. Laryngoscope. 2018 Aug;128(8):1898-1903. doi: 10.1002/lary.27201. Epub 2018 Apr 18. PMID 29668037
- [Background] Foote AG, Thibeault SL. Sensory Innervation of the Larynx and the Search for Mucosal Mechanoreceptors. J Speech Lang Hear Res. 2021 Feb 17;64(2):371-391. doi: 10.1044/2020_JSLHR-20-00350. Epub 2021 Jan 19. PMID 33465318
- [Background] Strohl MP, Chang JL, Dwyer CD, Young VN, Rosen CA, Cheung SW. Laryngeal Adductor Reflex Movement Latency Following Tactile Stimulation. Otolaryngol Head Neck Surg. 2022 Apr;166(4):720-726. doi: 10.1177/01945998211025517. Epub 2021 Jul 13. PMID 34253075
- [Background] Strohl MP, David AP, Dwyer CD, Rosen CA, Young VN, Chang JL, Cheung SW. Aesthesiometer-Based Testing for Laryngopharyngeal Hyposensitivity. Laryngoscope. 2022 Jan;132(1):163-168. doi: 10.1002/lary.29761. Epub 2021 Jul 20. PMID 34289117
- [Background] Strohl MP, Young VN, Dwyer CD, Bhutada A, Crawford E, Chang JL, Rosen CA, Cheung SW. Novel Adaptation of a Validated Tactile Aesthesiometer to Evaluate Laryngopharyngeal Sensation. Laryngoscope. 2021 Jun;131(6):1324-1331. doi: 10.1002/lary.28947. Epub 2020 Jul 31. PMID 32735711
- [Background] Aviv JE, Martin JH, Kim T, Sacco RL, Thomson JE, Diamond B, Close LG. Laryngopharyngeal sensory discrimination testing and the laryngeal adductor reflex. Ann Otol Rhinol Laryngol. 1999 Aug;108(8):725-30. doi: 10.1177/000348949910800802. PMID 10453777
- [Background] Shembel AC, Rosen CA, Zullo TG, Gartner-Schmidt JL. Development and validation of the cough severity index: a severity index for chronic cough related to the upper airway. Laryngoscope. 2013 Aug;123(8):1931-6. doi: 10.1002/lary.23916. Epub 2013 Jun 4. PMID 23737389
- [Background] DiBardino DM, Lanfranco AR, Haas AR. Bronchoscopic Cryotherapy. Clinical Applications of the Cryoprobe, Cryospray, and Cryoadhesion. Ann Am Thorac Soc. 2016 Aug;13(8):1405-15. doi: 10.1513/AnnalsATS.201601-062FR. PMID 27268274